CLINICAL TRIAL: NCT06075966
Title: The Study of INTRA Spine Non Fusion Technique in the Treatment of Lumbar Degenerative Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INTRA Spine
Record Dates: First submitted 2023-09-16; First posted 2023-10-10 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Degenerative Disease
Keywords: INTRA Spine system; dynamic stabilization; non-fusion; Lumbar degeneration; Lumbar range of motion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-fusion group (Experimental): Patients who have undergone the INTRA-Spine dynamic stabilization system insertion surgery for lumbar spondylosis and have complete follow-up data and meet the standards completed at the First Affiliated Hospital of Shandong First Medical University.
  Interventions: Other: Non-fusion group; Other: Fusion group
- Fusion group (Active Comparator): Patients who have undergone lumbar spine fusion surgery due to lumbar spondylosis and meet the standards and have complete follow-up data completed at the First Affiliated Hospital of Shandong First Medical University.
  Interventions: Other: Non-fusion group; Other: Fusion group

INTERVENTIONS:
Other: Non-fusion group — Patients who have undergone the INTRA-Spine dynamic stabilization system insertion surgery for lumbar spondylosis and have complete follow-up data and meet the standards completed at the First Affiliated Hospital of Shandong First Medical University.
Other: Fusion group — Patients who have undergone lumbar spine fusion surgery due to lumbar spondylosis and meet the standards and have complete follow-up data completed at the First Affiliated Hospital of Shandong First Medical University

SUMMARY:
Lumbar degenerative diseases such as lumbar disc herniation (LDH) and lumbar spinal stenosis (LSSS) are common and frequently encountered in orthopaedics. With the acceleration of the aging process of society, their incidence rate increases year by year. At present, conservative treatment is the preferred choice for this type of disease, and surgical treatment is feasible in cases where conservative treatment is ineffective. The main surgical methods include simple laminectomy and nucleus pulposus removal, intervertebral fusion and internal fixation, intervertebral disc replacement, and non fusion surgery. Simple nucleus pulposus removal surgery has drawbacks such as loss of intervertebral height and foramen height, which can affect spinal stability; Intervertebral fusion and internal fixation surgery has the problem of accelerating adjacent segment degeneration; The current therapeutic effect of lumbar disc replacement is not yet clear, and the technology is not yet mature. In response to the shortcomings of the above surgical methods, the advancement of science and technology has driven the development of spinal surgery, and a new surgical concept has emerged - spinal non fusion fixation technology. The INTRA-Spine dynamic stability system between vertebral lamina is one of the non fusion technologies of the spine. The core concept of this technology is to provide dynamic fixation on the basis of sufficient decompression of nerves, with the rotation center located between the vertebral lamina, which is closer to the normal movement center of the lumbar spine. It simulates the normal physiological structure of the lumbar spine with minimal damage and trauma, and maximizes the preservation of surgical segment mobility while maintaining spinal stability, Reducing stress concentration in adjacent segments caused by local fusion, thereby reducing the acceleration of adjacent segment degeneration, theoretically has good clinical and imaging efficacy.

DETAILED DESCRIPTION:
Retrospective analysis of patients admitted to the Department of Orthopedic and Spinal Surgery of our hospital who underwent the INTRA Spine dynamic stabilization system and lumbar fusion technology for the treatment of lumbar degenerative diseases. General, clinical, and imaging data were collected before and 7 days, 6 months, and 12 months after surgery. The general information of the patient includes gender, age, course of disease, conservative treatment time, surgical time, nail/implant placement time, bleeding volume, and length of hospital stay; The clinical treatment effect was evaluated using the visual analogue VAS score for low back and leg pain, the Japanese Orthopedic Association's JOA score for evaluation of treatment, and the Oswestry Dysfunction Index questionnaire ODI score; The imaging data includes measuring the lateral position of the surgical segment and adjacent segments through lumbar lateral X-ray films, the Cobb angle, flexion and extension range of motion (ROM), intervertebral disc height, and intervertebral foramen height in the over extension and over flexion positions. The optimal measurement angle value is used, and each measurement data is measured three times and its mean is taken. Perform analysis of variance (intra group follow-up time) and t-test (inter group) on the obtained data using statistical software SPSS; Statistics and analysis of clinical efficacy and imaging manifestations.This clinical study has a funding of 50000 RMB.

ELIGIBILITY:
Inclusion Criteria:

* The patient's clinical manifestations, physical examination, and imaging data all support the diagnosis of degenerative lumbar spondylosis
* Those who have undergone strict and formal conservative treatment for at least 3 months before surgery and have no significant improvement in symptoms
* Preoperative imaging examination showed single responsible segment protrusion or protrusion leading to segment stenosis
* Surgeries are performed by the same chief surgeon.

Exclusion Criteria:

* Lumbar instability, lumbar spondylolisthesis above grade II
* Patients with severe osteoporosis, tuberculosis, or tumors
* Systemic diseases that affect surgical treatment and medication, such as heart disease, liver disease, and kidney disease
* Patients with mental illness, poor compliance, and inability to cooperate in completing follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS | 2 Years
  The visual analog scale (VAS) is used for pain assessment. It is widely used in clinical practice in China, and the basic method is to use a vernier ruler with a length of about 10cm, marked with 10 scales on one side, with both ends marked as "0" and "10" respectively. A score of 0 indicates painlessness, and a score of 10 represents the most severe pain that cannot be tolerated.
JOA | 2 Years
  The Japanese Orthopaedic Association Scores (JOA) is a neurological function scoring system recommended by the Japanese Orthopaedic Association, which includes four parts: upper limb motor function, lower limb motor function, sensory and bladder function, with a total score of 29 points. The lower the score, the more severe the neurological dysfunction.
Cobb angle of surgical space and adjacent space in neutral position, over extension and over flexion position | 2 Years
  Cobb angle of surgical space and adjacent space in neutral position, over extension and over flexion position

SECONDARY OUTCOMES:
ROM,range of motion | 2 Years
  range of motion
posterior disc height, PDH | 2 years
  posterior disc height
foraminal height ,FH | 2 years
  foraminal height

CONTACTS AND LOCATIONS:
Overall Officials: Hao-Xuan Zhang, Ph.D/MD, Study Chair — Shandong First Medical University
Locations (2):
- China (2):
  - Hao-Xuan Zhang, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT06075966/Prot_SAP_000.pdf